CLINICAL TRIAL: NCT00366626
Title: Alcohol Research Center Grant. Component #1: Naltrexone Effects on Alcohol Reactivity and Consumption, Evaluating the Genetic Variability of Naltrexone Response
Brief Title: Effectiveness of Naltrexone Versus Placebo to Reduce Craving for Alcohol With Evaluation of Genetic Variability.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50AA010761 (NIH)
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2012-11

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Alcoholism; Craving; Genetic
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. (Experimental): Naltrexone one capsule a day
  Interventions: Drug: Naltrexone
- 2 (Placebo Comparator): One capsule a day match to naltrexone
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Naltrexone (25 mg/day for days 1-2 and 50 mg/day for days 3-7)
  Other Names: ReVia
  Arms: 1.
Drug: Placebo — Placebo for 7 days matched to Naltrexone
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether naltrexone (an opiate blocking agent approved for the treatment of alcohol dependence) is more effective in the reduction of alcohol craving and drinking compared to placebo in individuals with particular genetic predisposition.

DETAILED DESCRIPTION:
About 300 non-treatment seeking alcoholics will be recruited through advertisement and paid for their participation. They will be assessed, subtyped for mu-opiate receptor and catechol-O-methyltransferase (COMT) allelic variants and 88 individuals (44 with the more common AA gene and 44 with either an AG or GG gene) will be randomly assigned to take either naltrexone (50 mg/day) or a matching placebo for 7 days. Since the val and met alleles of the catechol-O-methyltransferase (COMT) gene are each present in about 50% of the population they will be equally distributed by urn randomization to all opiate allele and treatment groups. After 5 days of natural drinking and one day of abstinence, subjects will undergo an alcohol cue-induced brain activity scan using well-established fMRI techniques on Day 6 of study drug. The following day all subjects will receive a standard dose (gender and weight corrected) of alcohol and be evaluated for alcohol reactivity (stimulation, sedation, intoxication, craving) over 40 minutes. They then will be allowed to consume up to 8 mini-drinks over a 2-hour period. Afterwards all subjects will receive educational/motivational counseling regarding their alcohol use and its effects. Referral for treatment will be offered.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 21-65. 2. Meets the DSM IV criterion for current alcohol dependence including "loss of control over drinking" (criterion 4) but does not necessarily have signs of physiologic dependence as expressed in criterion for tolerance development (criterion 1) and withdrawal symptoms or use to avoid withdrawal symptoms (criterion 2).

  3. Drinks hard liquor/spirits and does not have aversion to this form of alcohol.

  4. Drinks alone (not in the presence of others) some of the time (to maximize the potential of drinking in the bar lab where a subject will not be in the company of others).

  5. Currently is not engaged in, and does not want treatment for, alcohol related problems.

  6. Able to read and understand questionnaires and informed consent. 7. Lives within 50 miles of the study site. 8. Able to maintain abstinence for two days (without the aid of detox medications) as determined by self-report and breathalyzer measurements.

Inclusion for fMRI imaging sub-study (see methodology section for rationale):

1. Does not have metal objects in the head/neck.
2. Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.

Exclusion Criteria:

* 1. Currently meets DSM-IV criteria for any other psychoactive substance dependence disorder.

  2. History of opiate abuse or a positive urine drug screen for opiates. 3. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days as evidenced by self-report and urine drug screen. For marijuana - no use within the last seven days.

  4. Meets DSM-IV criteria for current axis I disorders of major depression, panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, bipolar affective disorder, schizophrenia, dissociative disorders and eating disorders, any other psychotic disorder or an organic mental disorder.

  5. Has current suicidal ideation or homicidal ideation. 6. Need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications.

  7. Current use of disulfiram, naltrexone, or acamprosate. 8. Clinically significant medical problems such as, cardiovascular, renal, gastrointestinal, or endocrine problems that would impair participation or limit medication ingestion.

  9. Past history of alcohol related medical illness such as gastrointestinal bleeding, pancreatitis, peptic ulcer, hepatic cirrhosis or alcoholic hepatitis.

  10. Hepatocellular disease indicated by elevations of SGPT Alanine transaminase(ALT) or SGOT Aspartate transaminase(AST) greater than 3 times normal at screening.

  11. Females of child-bearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.

  12. Has current charges pending for a violent crime (not including DUI related offenses).

  13. Does not have a stable living situation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Anton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- · Center for Drug and Alcohol Programs,· Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Anton RF, Voronin KK, Randall PK, Myrick H, Tiffany A. Naltrexone modification of drinking effects in a subacute treatment and bar-lab paradigm: influence of OPRM1 and dopamine transporter (SLC6A3) genes. Alcohol Clin Exp Res. 2012 Nov;36(11):2000-7. doi: 10.1111/j.1530-0277.2012.01807.x. Epub 2012 May 2. PMID 22551036

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 38 | 45
Completed | 38 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 38 | 45 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 45 | 83
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (10) | 26 (10) | 28 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 25 | 29 | 54
Region of Enrollment [Number; unit: participants]
  United States | 38 | 45 | 83

OUTCOME MEASURES:

1. Primary Outcome: "Natural" Alcohol Consumption Period; Average Number of Drinks Per Day Consumed During the 5 Day Natural (Usual Environment) Drinking Observation Period
Time Frame: treatment days 1 - 5
Population: All subjects who were randomized.
Measure: Mean (Standard Deviation); unit: Drinks per day
Groups:
- Naltrexone (asn40asn): Subjects with asn40asn OPRM1 SNP who got Naltrexone during he study
- Naltrexone (asp40): Subjects with asp40 OPRM1 SNP who got Naltrexone during he study
- Placebo (asn40asn ): Subjects with asn40asn OPRM1 SNP who got Placebo during he study
- Placebo (asp40): Subjects with asp40 OPRM1 SNP who got Placebo during he study
Arm/Group | Naltrexone (asn40asn) | Naltrexone (asp40) | Placebo (asn40asn ) | Placebo (asp40)
Number analyzed (Participants) | 19 | 19 | 21 | 24
Drinks per day | 4.7 (1.8) | 5.7 (3.2) | 6.2 (3.4) | 6.3 (3.7)
Statistical Analysis 1: Comparison: Naltrexone (asn40asn) vs Naltrexone (asp40) vs Placebo (asn40asn ) vs Placebo (asp40); This was a 2 gene (asn40asn vs 40asp) by two medication (naltrexone vs placebo) design. The main hypothesis was that the effect of naltrexone (mean naltrexone drinking - placebo drinking) would be greater in the 40asp subjects than in the asn40asn subjects. Thus the null hypothesis there would be no gene by medication interaction. The mean difference above is then the difference in the size of the naltrexone effect in the two genotypes, equivalent to the interaction; Test type: Superiority or Other; p = 0.51, ANOVA; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-1.85 to 3.69], Standard Deviation 6.32

2. Primary Outcome: Limited Access Alcohol Consumption Paradigm; Total Number of Drinks Consumed
Description: Subjects were allowed to drink up to 8 alcohol drinks during 2 hours observation period being in bar/laboratory settings vs to get $2 per each not consumed drink.
Time Frame: On day 7 of treatment during limited access alcohol consuption in the bar/laboratory
Population: All subjects who were randomized.
Measure: Mean (Standard Deviation); unit: Total number of drinks consumed
Arm/Group | Naltrexone (asn40asn) | Naltrexone (asp40) | Placebo (asn40asn ) | Placebo (asp40)
Number analyzed (Participants) | 19 | 19 | 21 | 24
Total number of drinks consumed | 3.0 (2.9) | 3.8 (3.1) | 3.8 (2.8) | 3.1 (3.3)
Statistical Analysis 1: Comparison: Naltrexone (asn40asn) vs Naltrexone (asp40) vs Placebo (asn40asn ) vs Placebo (asp40); This was a 2 gene (asn40asn vs 40asp) by 2 medication (naltrexone vs. placebo)interaction analysis. The main hypothesis was that subjects who had 40asp OPRM1 allele would a greater naltrexone effect on drinking (Placebo - Naltrexxone) than the asn40asn subjects. Thus the null hypothesis was the gene by medication interaction; Test type: Superiority or Other; p = 0.28, ANOVA; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [-1.22 to 4.11], Standard Deviation 6.1

ADVERSE EVENTS:
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/45
Other Adverse Events (participants affected / at risk) | 0/38 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes